CLINICAL TRIAL: NCT00842556
Title: Pharmacokinetic Drug Interaction Study of Dapagliflozin and Glimepiride or Sitagliptin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MB102-037
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; glimepiride; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dapagliflozin (Active Comparator)
  Interventions: Drug: Dapagliflozin
- Glimepiride (Active Comparator)
  Interventions: Drug: Glimepiride
- Dapagliflozin + Glimepiride (Active Comparator)
  Interventions: Drug: Dapagliflozin; Drug: Glimepiride
- Sitagliptin (Active Comparator)
  Interventions: Drug: Sitagliptin
- Dapagliflozin + Sitagliptin (Active Comparator)
  Interventions: Drug: Dapagliflozin; Drug: Sitagliptin

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 20 mg, Single Dose
  Other Names: BMS-512148
  Arms: Dapagliflozin; Dapagliflozin + Glimepiride; Dapagliflozin + Sitagliptin
Drug: Glimepiride — Tablets, Oral, 4 mg, Single Dose
  Other Names: Amaryl
  Arms: Dapagliflozin + Glimepiride; Glimepiride
Drug: Sitagliptin — Tablets, Oral, 100 mg, Single Dose
  Other Names: Januvia
  Arms: Dapagliflozin + Sitagliptin; Sitagliptin

SUMMARY:
To assess the effect of glimepiride on the PK of dapagliflozin and the effect of dapagliflozin on the PK of glimepiride, when co-administered in healthy subjects (Phase A) and to assess the effect of sitagliptin on the PK of dapagliflozin and the effect of dapagliflozin on the PK of sitagliptin, when co-administered in healthy subjects (Phase B)

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Body mass index (BMI) of 18 to 32 kg/m2, inclusive BMI = weight (kg)/[height(m)]2

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 12 weeks after the last dose of investigational product
* Abnormal liver functions tests (ALT, AST or total bilirubin > 10% above ULN)
* History of chronic or recurrent UTI (defined as 3 occurrences per year) or UTI in the past 3 months
* History of allergy to SGLT@ inhibitors, DPP$ inhibitors or sulfonylurea or related compounds
* Prior exposure to dapagliflozin, sitagliptin and glimepiride within 3 months of Day -1
* History of recurrent (defined as 3 occurrences per year) or recent vulvovaginal mycotic infections

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Exposure to the investigational drug will be measured to compare with and without the co-administration of other drugs | 72 hours after dosing

SECONDARY OUTCOMES:
To assess the safety and tolerability in healthy subjects | 15 time points up to 72 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Austin, Texas, United States

REFERENCES:
- See also: MB102-037_Redacted _CSR _synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3643&filename=MB102-037_Redacted%20_CSR%20_synopsis.pdf